CLINICAL TRIAL: NCT06138171
Title: Psychological Layers of Nociplastic Pain: Cluster Analysis of The Role of Personality Traits, Defence Mechanisms, Central Sensitization, and Childhood Traumatic Experiences in Patients With Chronic Migraine, Fibromyalgia, and Vulvodynia
Brief Title: Personality, Defences, Central Sensitization, and Trauma in Women With Chronic Migraine, Fibromyalgia, and Vulvodynia
Acronym: PSYCHOFIBRO
Status: Completed | Type: Observational
Sponsor: University of Roma La Sapienza (Other)
Collaborators: University of Milan (Other); Pavia IRCCS Mondino di Pavia (Unknown); Azienda Policlinico Umberto I (Other)
Responsible Party: Principal Investigator, Federica Galli, Professore Associato (Associate Professor), University of Roma La Sapienza
Other Study IDs: 0001979
Record Dates: First submitted 2023-11-07; First posted 2023-11-18 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Fibromyalgia; Chronic Migraine, Headache; Vulvodynia
Keywords: central sensitivity; traumatic childhood experiences; mental pain; environmental sensitivity; defense mechanisms
MeSH Terms: conditions — Fibromyalgia; Headache; Vulvodynia | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Fibromyalgia - FM: Cohort of women diagnosed with FM recruited consecutively in the clinical department following the criteria:
  * age range 18-65 years
  * education > 5 years
  * diagnosis of FM according to Wolfe, 2016
  Exclusion criteria
  * severe psychiatric disorders and/or cognitive impairment
  * difficulties in comprehension/expression in Italian
  * history of other chronic pain disorder(s)
  * history of other neurological disorders besides migraine
  Interventions: Other: Psychological self-reported measures assesment (questionnaire)
- Chronic migraine - CM: Cohort of women diagnosed with CM recruited consecutively in the clinical department following the criteria:
  * age range 18-65 years
  * education > 5 years
  * diagnosis of CM according to Olesen, 2017
  Exclusion criteria
  * severe psychiatric disorders and/or cognitive impairment
  * difficulties in comprehension/expression in Italian
  * history of other chronic pain disorder(s)
  * history of other neurological disorders besides migraine
  Interventions: Other: Psychological self-reported measures assesment (questionnaire)
- Vulvodynia - VU: Cohort of women diagnosed with VU recruited consecutively in the clinical department following the criteria:
  * age range 18-65 years
  * education > 5 years
  * diagnosis of VU according to Bornstein et al., 2016
  Exclusion criteria
  * severe psychiatric disorders and/or cognitive impairment
  * difficulties in comprehension/expression in Italian
  * history of other chronic pain disorder(s)
  * history of other neurological disorders besides migraine
  Interventions: Other: Psychological self-reported measures assesment (questionnaire)
- Control group (no chronic pain condition): Cohort of women recruited consecutively from the general population with the following criteria:
  * age range 18-65 years
  * education > 5 years
  * no previous diagnosis of chronic pain conditions
  Exclusion criteria
  * severe psychiatric disorders and/or cognitive impairment
  * difficulties in comprehension/expression in Italian
  * history of other chronic pain disorder(s)
  * history of other neurological disorders
  Interventions: Other: Psychological self-reported measures assesment (questionnaire)

INTERVENTIONS:
Other: Psychological self-reported measures assesment (questionnaire) — The study involves the administration of a protocol of self-report questionnaires consisting of two parts: the main (about 25 minutes for the administration) and the optional one (additional 20 minutes). This decision stems from the realization of the length of the protocol, to increase the collection of data in pursuit of the main objective of the study (cluster analysis).

SUMMARY:
Chronic pain (CP) is a substantial healthcare challenge with considerable economic costs. Recently, the term Nociplastic Pain (NP) has been introduced as a third descriptor of mechanisms related to CP. NP describes conditions that arise from altered nociception despite no clear evidence of actual or threatened tissue damage. It represents a new way of describing somatoform painful conditions, originating from altered central-nervous pathways (e.g., central sensitization) and with the important involvement of clinical psychological factors. Among nociplastic chronic syndromes have been included fibromyalgia (FM), chronic migraine (CM) and vulvodynia (VU). These chronic pain disorders have been usually studied separately, although the high comorbidity rates. Many studies evidenced the role of psychosocial variables in the onset and maintenance of the burden related to these conditions. Among them, personality traits, defense mechanisms, central sensitization, and childhood traumatic experiences may play a pivotal role in the onset of the NP. The first aim of this study is to highlight possible psychosocial clusters of variables that are specific for each condition (FM, CM, and VU). A second aim, to improve the tailored psychological treatment devoted to these conditions, is to explore the association between FM, CM, and VU with depression, anxiety, somatization, quality of life, alexithymia, social support, sexual satisfaction, and functioning. This will make it possible to identify specifically for each condition the areas of greatest interest that can be investigated and treated in clinical intervention. To identify specific descriptors, NP conditions will be compared with a control group of subjects reporting other types of CP (e.g., knee arthrosis, rheumatoid arthritis). The study involves the collection of data from a self-administered questionnaire in several Italian centers specializing in the above-mentioned clinical conditions under the guidance of the research team of the Department of Dynamic and Clinical Psychology and Health Studies, PI Professor Federica Galli.

DETAILED DESCRIPTION:
Chronic pain (CP), defined as pain lasting more than 3 months, is a substantial healthcare challenge. Prevalence rates of CP are between 11% and 40% (Dahlhamer et al., 2018; Fayaz et al., 2016). CP prevalence increases with age, is greater among females, and among people with lower socioeconomic status (Tsang et al., 2008; Pergolizzi et al., 2013). CP affects relationships and self-esteem, and is associated with higher divorce and suicide rates, and an increased risk of substance abuse (Tang et al., 2016; Fitzcharles et al., 2021), psychopathology (Katz et al., 2015) and risk of medication overuse (Westergaard et al., 2015). The causes of CP are still poorly understood. Recently, the International Association for the Study of Pain (IASP, 2017) has proposed that three subtypes of CP may be differentiated based on unique causal mechanisms: nociceptive, neuropathic, and nociplastic.

Nociplastic Pain (NP) is a new descriptor of CP and includes conditions that arise from altered nociception despite no clear evidence of actual or threatened tissue damage. NP should be viewed as an overarching term that can be applied to a diverse range of clinical conditions that share common neurophysiological mechanisms, involving various organ systems (Galli, 2023). Among nociplastic chronic syndromes have been included chronic migraine, fibromyalgia, and vulvodynia (Bergeron et al., 2020; Fitzcharles et al., 2021). NP is usually accompanied by other central nervous system-associated symptoms with a close link with clinical psychological factors: general symptoms (e.g., fatigue and cognitive problems), temperamental characteristics (e.g., hypersensitivity to environmental stimuli) and psychological symptoms (e.g., anxiety/depression) (Fitzcharles et al., 2021). Many emotional states, such as depression and anxiety, and emotional processes, such as emotional awareness and regulation, may influence the presence and severity of NP (Aaron et al., 2020; Lumley et al., 2021), opening to the importance of a psychological assessment for diagnosis and psychological interventions. The concept of NP opens a new framework for understanding the co-occurrence of different chronic disorders and the role of related psychological factors. Comorbid chronic disorders may be the expression of shared pathophysiological mechanisms, with etiological and psychological features differentiating them by "pure" forms of the same disease. The comorbid association of migraine, fibromyalgia, and vulvodynia, and the well-known link with clinical psychological factors (e.g., early traumatic events, anxiety and depression, alexithymia, dissociation, etc.) is quite established (Bergeron et al., 2020; Fitzcharles et al., 2021). However, these chronic pain disorders have been usually studied as separate diseases. On the one hand, this research project wants to observe the common basis of these chronic pain disorders, which can be traced back to central sensitization mechanisms, the influence of early adverse events, and other psychological factors, and on the other hand it wants to observe the psychosocial peculiarities of each assessed condition (fibromyalgia, migraine, and vulvodynia) for tailored treatment purposes.

CHRONIC MIGRAINE (CM) Migraine affects ~15% of the general population globally and is typically characterized by recurring, often highly disabling attacks of severe headache, nausea, vomiting, super- sensitivity to light and sound, and other variable physical, mental, and psychological signs and symptoms, lasting for 4-72 h (Ferrari et al., 2022). Migraine is listed by The Global Burden of Disease Study as the third most disabling disease worldwide (Vos et al., 2012). Most patients have episodic migraine, although some patients develop CM (the presence of ≥15 headache days per month). The 1- year prevalence of migraine is 8-15% worldwide, but is highly dependent on age, sex, and migraine subtype (Ferrari et al., 2015). Migraine is 40-60% determined by genetic factors and for the remainder by non- genetic risk- modulating and trigger factors. Although a progressive increase of the attack frequency can occur spontaneously, it is often aggravated and/or induced by overuse of acute headache medications and/or caffeine. Risk factors for migraine progression toward CM include high headache frequency, high headache-related disability, obesity, allodynia, anxiety, and depression (Ferrari et al., 2022). Comorbid migraine and anxiety/depression are common in the general population, but the mechanism(s) supporting the comorbidity are still unknown. Overall, there seems to be a bidirectional relationship between migraine and depression, and a shared pathophysiological mechanism has been recently outlined (Karsan & Goadsby, 2021). Indeed, in cohort studies, the risk of incident migraine in persons with existing major depression was threefold higher than in persons without depression, and incident major depression in persons with pre- existing migraine was more than fivefold higher than in persons without migraine history (Modgill et al., 2011). Comorbid anxiety/depression increases the risk of migraine chronification (Guidetti et al., 1998; Tietjen et al., 2007). However, there is no evidence that treating depression or anxiety mitigates migraine (Ferrari et al., 2022). Other psychological factors have been linked to migraine over time, as the case of alexithymia (Galli et al., 2017, Bottiroli et al., 2018), traumatic events (Bottiroli et al., 2019; Stensland et al., 2013), early episodes of maltreatment (Tietjen et al., 2016), personality characteristics (Bottiroli et al., 2016; 2021; Galli et al., 2019).

FIBROMYALGIA (FM) FM is a chronic syndrome characterized by widespread musculoskeletal pain associated with fatigue, nonrestorative sleep, and cognitive deficits (Wolfe et al., 2016) with high incidence among women (Branco et al., 2010). The prevalence of CP comorbidities among FM patients was also high ranging from 39% to 76% (with headache and irritable bowel syndrome that were the most prevalent). Although a central sensitization phenomenon seems to play a central role in FM (Arnold et al., 2016), the etiopathology of FM remains unknown (Thieme et al., 2017). For these reasons, researchers have proposed a biopsychosocial model of interacting variables that can activate and exacerbate FM symptoms (Sommer et al., 2012). FM patients experience excessive levels of psychological distress: 20-80% experience anxiety and 13-64% experience depression (Galvez-Sánchez et al., 2019). A recent systematic review on comorbidities in FM (Kleykamp et al., 2021) found that the most prevalent comorbidity across all studies reviewed was depression/major depressive disorder with over half of the patients included having this diagnosis in their lifetime. Another interesting personality construct involved in FM is 'distressed' personality (van Middendorp et al., 2016). Moreover, nearly one-third of FM patients had current or lifetime bipolar disorder, panic disorder, or post-traumatic stress disorder. Specifically, among environmental factors, stressful life events have been considered (Nakamura et al., 2014). Trauma and major life stress are unlikely to cause FM per se. In genetically susceptible persons, it is likely that early trauma and prolonged stress in adulthood will influence brain modulatory circuitry of both pain and emotions (Crofford, 2007; Schweinhardt et al., 2008) that could explain the increased pain responses and symptoms of patients with FM. Traumatic events have been shown to influence pain severity as well (Bote et al., 2013). Several theoretical models have suggested that some personality characteristics lead to a worse response to stressors and adjustment to diseases in people with CP, such as FM (Naylor et al., 2017; Galvez-Sánchez et al., 2019). A minority of studies have focused on the detection of personality disorders associated with FM (Attademo & Bernardini, 2018). In general, previous studies found a high prevalence of avoidance (41.4%), obsessive-compulsive (33.1%) and borderline personality disorder (5.2-27.4%) in FM (Thieme et al., 2004; Uguz et al., 2010; Gumà-Uriel et al., 2016). In recent years, many studies on FM have reported a high prevalence of alexithymia (15-20%) (Di Tella et al., 2017; Marchi et al., 2019; Atzeni et al., 2019).

VULVODYNIA Vulvodynia is a condition that occurs in 8-10% of women of all ages (Arnold et al., 2007; Harlow et al., 2014) and is characterized by localized pain in the vulva, either spontaneous or upon touch, and can occur during sexual and/or non-sexual situations (Bergeron et al., 2020). Vulvodynia has a negative effect on the quality of life of women and their partners and imposes a profound personal and social economic burden. The diagnosis is established through a careful history and pelvic examination, including the cotton swab test, based on persistent vulvar pain lasting more than 3 months without an identifiable cause and with several potential associated factors. These include musculoskeletal and neurological factors, comorbid pain syndromes (such as fibromyalgia, chronic migraine, and irritable bowel syndrome) and psychosocial factors (Reed et al., 2012; Wesselmann et al., 2014; Bergeron et al., 2020). Current literature suggests that the onset and maintenance of vulvodynia likely involves a complex interplay of peripheral and central pain mechanisms, pelvic floor muscle and autonomic dysfunction, anxiety, depression, and adverse childhood events, as well as cognitive-affective, behavioral, and interpersonal factors (Bergeron et al., 2020). Vulvodynia has traditionally been conceptualized in a dualistic manner, arising from either physical factors or psychological and sexual difficulties, although research contrary to this concept and other hypotheses suggest that these two perspectives should be combined. Therefore, future studies should move in this direction, seeking to identify specific pathophysiological mechanisms within the framework of a biopsychosocial model. Indeed, a more recent theorization has focused on an integrated model that considers the interdependence of biopsychosocial factors in vulvodynia and associated disorders, in which medical and psychosocial mechanisms are considered to contribute to the onset, chronicization and exacerbation of pain and associated difficulties (Bergeron et al., 2011). The neurophysiology of vulvodynia is multifaceted. It is characterized by both peripheral and central sensory abnormalities (Wesselmann et al., 2014; Pukall et al., 2016). Furthermore, increased sensitivity to different sensory modalities at extragenital sites has been demonstrated in women with vulvodynia (Giesecke et al., 2004; Foster et al., 2005; Sutton et al., 2015), suggesting central sensitization. This central sensitization could explain the observation of overlapping chronic pain conditions in women with vulvodynia, which need further investigation to be better understood.

PSYCHOLOGICAL FACTORS ASSOCIATED TO NP As the investigators have already pointed out separately for the three pathological conditions (chronic migraine, fibromyalgia, and vulvodynia), there is evidence that factors such as personality traits, defense mechanisms, central sensitization, and childhood traumatic experiences may contribute significantly to the genesis of these disorders through a process of central sensitization of pain pathways. Central sensitization (CS) is defined as increased responsiveness of nociceptive neurons in the central nervous system to their normal or subthreshold afferent input according to the IASP - International Association for the Study of Pain (Arendt-Nielsen et al., 2018). A sensitized nervous system has been considered one of the most important mechanisms involved in NP (Cohen, 2022). CS plays a role in fibromyalgia, in which alteration of central nociceptive processing occurs and pain can be worsened by psychological factors (Sluka & Clauw, 2016). In migraine, CS may contribute to acute allodynia and headache chronification (De Tommaso & Sciruicchio, 2016). Furthermore, in migraine CS may play a role in trigeminal nerve activation and cortical spreading depression (De Tommaso & Sciruicchio, 2016). It has been suggested that migraine may be considered as a brain state of altered excitability and a disorder of sensory processing (Goadsby et al., 2017), encompassing additional symptoms as fatigue and mood disorders (Karsan & Goadsby, 2021). Structural and functional MRI studies in women with provoked vulvar or distant/extra- genital pain have supported a role of central sensitization and dysregulation of endogenous pain modulatory systems in the central nervous system in the pathophysiology of vulvodynia (Bergeron et al., 2020).

In the process of central sensitization, psychological factors such as traumatic events in childhood, the development of specific personality expressions (traits), and the use of different forms of defense mechanisms also play a role. No study to our knowledge has yet tried to identify specific clusters of psychological factors (personality traits, defense mechanisms, central sensitization, and childhood traumatic experiences) capable of characterizing or differentiating between the different pathologies expressed by a NP.

In addition to this, the study of psychosocial factors associated with the experience of such pathologies or possible emerging clusters such as depression, anxiety, somatization, quality of life, alexithymia, social support, sexual satisfaction, and functioning. This will make it possible to identify specifically for each condition the areas of greatest interest that can be investigated and treated in clinical intervention tailored to the person.

Aims To highlight possible psychosocial clusters of variables that are specific to the onset and maintenance for each condition (FM, CM, and VU). Specifically, the observation of possible clusters will be made based on variables such as personality traits, defense mechanisms, central sensitization, and childhood traumatic experiences. The hypothesis is that specific psychological factors (clusters of high number of early traumatic events, high levels of central sensitization, and specific traits and defense mechanisms) characterize FM, CM, and VU groups compared to controls.

ELIGIBILITY:
Inclusion criteria:

* age range 18-65 years
* education > 5 years
* diagnosis of FM according to Wolfe, 2016
* diagnosis of CM according to Olesen, 2017
* diagnosis of VU according to Bornstein et al., 2016

Exclusion criteria

* severe psychiatric disorders and/or cognitive impairment
* difficulties in comprehension/expression in Italian
* history of other chronic pain disorder(s)
* history of other neurological disorders besides migraine

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study involves the collection of data from a self-administered questionnaire in several Italian centers specializing in the above-mentioned clinical conditions. The four centers involved in the recruitment of the participants will be the Università di Milano IRCCS Sant'Ambrogio Galeazzi under the haed of Prof. Sarzi-Puttini and Dott. Valeria Giorgi, the IRCCS Mondino di Pavia under the head of Prof. Cristina Tassorelli and Prof. Sara Bottiroli, The Policlino San Matteo of Paviaunder the head of Prof. Rossella Nappi and Dott. Lara Tiranini, and the Policlinico Umberto I of Sapienza University of Rome under the head of Dott. Cristina Iannuccelli.
  Questionaires will be accessible online through a web survey available on the Google.forms platform. Participants will provide an informed consent before accessing the survey, and the questionnaire will be anonymous with no remuneration provided.
Sampling Method: Non-Probability Sample
Enrollment: 1006 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Central sensitivity index | Day 0
  Central Sensitivity Inventory (CSI) (Chiarotto et al., 2018). Range scores go from 0 to 100, with higher scores indicating worse conditions.
Traumatic experiences index | Day 0
  Traumatic Experiences Checklist (TEC) (Nijenhuis et al., 2002). Range scores go from 0 to 29, with higher scores indicating more traumatic experiences in life.
Personality traits | Day 0
  PID-5 Short form (Thimm et al., 2016). Range scores go from 0 to 75, with higher scores indicating higher presence of disfunctional personality traits
Defense mechanisms | Day 0
  Defense Mechanism Rating Scales - DMRS-SR-30 (Di Giuseppe et al., 2020). Range scores go from 3.5 to 7, with higher scores indicating more consistent use of defense mechanisms.
Mental pain | Day 0
  Mental Pain Questionnaire (Svicher et al., 2019). Range scores go from 0 to 10, with higher scores indicating worse conditions.
Environmental sensitivity | Day 0
  Highly Sensitive Person Scale (HSP-12) (Aron & Aron, 1997; Lionetti et al., 2018). Range scores go from 1 to 7, with higher scores indicating worse conditions.

SECONDARY OUTCOMES:
Presence and intensity of psychological symptoms of depression, anxiety and psychosomaitcs | Day 0
  Brief Symptom Inventory (BSI-18) (Franke et al., 2017) Range scores go from 0 to 4, with higher scores indicating worse conditions.
Physical and Psychological Quality of life index | Day 0
  SF-12 - Quality of Life Assessment (Apolone et al., 2001). Range scores go from 0 to 100, with higher scores indicating better quality of life.
Alexithymic traits | Day 0
  Toronto Alexithymia Scale (TAS-20) (Bagby et al., 1994). Range scores go from 20 to 100, with higher scores indicating higher alexithymic traits.
Percieved Social Support | Day 0
  SPQ - Social Support Questionnaire (SPQ) (van der Lugt et al., 2012). Range scores go from 0 to 24, with higher scores indicating higher support received by social network.
Sexual Satisfaction | Day 0
  Sexual Satisfaction Scale (SSS) - Short form) (Meston & Trapnell, 2005). Range scores go from 6 to 30, with higher scores indicating higher level of sexual satisfaction.
gentipolvic pain | Day 0
  Short Form McGill Questionnaire (SF-MGQ) - Adapted for genito-pelvic pain (Melzack & Raja, 2005). Range scores go from 0 to 83, with higher scores indicating more genital pain.
Sexual Functioning | Day 0
  Female Sexual Function Index (FSFI) (Rosen et al., 2000). Range scores go from 2.6 to 36, with higher scores indicating better sexual health.

CONTACTS AND LOCATIONS:
Overall Officials: Federica M Galli, AP, Principal Investigator — University of Roma La Sapienza
Locations (1):
- Sapienza University of Rome, Department of Dynamic and Clinical Psychology and Health Studies, Rome, Italy

IPD SHARING:
Plan to Share IPD: Undecided
We are planning to upload data on dataverse after the end of collection phase

REFERENCES:
- [Background] Apolone, G., Mosconi, P., Quattrociocchi, L., Gianicolo, E., Groth, N., & Ware Jr, J. E. (2001). Questionario sullo stato di salute SF-12 [Health Status Questionnaire SF-12]. Milano, Italia: Istituto di Ricerche farmacologiche Mario Negri.
- [Background] Arendt-Nielsen L, Morlion B, Perrot S, Dahan A, Dickenson A, Kress HG, Wells C, Bouhassira D, Drewes AM. Assessment and manifestation of central sensitisation across different chronic pain conditions. Eur J Pain. 2018 Feb;22(2):216-241. doi: 10.1002/ejp.1140. Epub 2017 Nov 5. PMID 29105941
- [Background] Arnold LD, Bachmann GA, Rosen R, Rhoads GG. Assessment of vulvodynia symptoms in a sample of US women: a prevalence survey with a nested case control study. Am J Obstet Gynecol. 2007 Feb;196(2):128.e1-6. doi: 10.1016/j.ajog.2006.07.047. PMID 17306651
- [Background] Arnold LM, Gebke KB, Choy EH. Fibromyalgia: management strategies for primary care providers. Int J Clin Pract. 2016 Feb;70(2):99-112. doi: 10.1111/ijcp.12757. PMID 26817567
- [Background] Aron EN, Aron A. Sensory-processing sensitivity and its relation to introversion and emotionality. J Pers Soc Psychol. 1997 Aug;73(2):345-68. doi: 10.1037//0022-3514.73.2.345. PMID 9248053
- [Background] Attademo L, Bernardini F. Prevalence of personality disorders in patients with fibromyalgia: a brief review. Prim Health Care Res Dev. 2018 Sep;19(5):523-528. doi: 10.1017/S1463423617000871. Epub 2017 Dec 22. PMID 29268809
- [Background] Atzeni F, Talotta R, Masala IF, Giacomelli C, Conversano C, Nucera V, Lucchino B, Iannuccelli C, Di Franco M, Bazzichi L. One year in review 2019: fibromyalgia. Clin Exp Rheumatol. 2019 Jan-Feb;37 Suppl 116(1):3-10. Epub 2019 Feb 6. PMID 30747097
- [Background] Bagby RM, Taylor GJ, Parker JD. The Twenty-item Toronto Alexithymia Scale--II. Convergent, discriminant, and concurrent validity. J Psychosom Res. 1994 Jan;38(1):33-40. doi: 10.1016/0022-3999(94)90006-x. PMID 8126688
- [Background] Bergeron S, Reed BD, Wesselmann U, Bohm-Starke N. Vulvodynia. Nat Rev Dis Primers. 2020 Apr 30;6(1):36. doi: 10.1038/s41572-020-0164-2. PMID 32355269
- [Background] Bergeron S, Rosen NO, Morin M. Genital pain in women: Beyond interference with intercourse. Pain. 2011 Jun;152(6):1223-1225. doi: 10.1016/j.pain.2011.01.035. Epub 2011 Feb 15. No abstract available. PMID 21324589
- [Background] Bornstein J, Goldstein AT, Stockdale CK, Bergeron S, Pukall C, Zolnoun D, Coady D; consensus vulvar pain terminology committee of the International Society for the Study of Vulvovaginal Disease (ISSVD), the International Society for the Study of Women's Sexual Health (ISSWSH), and the International Pelvic Pain Society (IPPS). 2015 ISSVD, ISSWSH and IPPS Consensus Terminology and Classification of Persistent Vulvar Pain and Vulvodynia. Obstet Gynecol. 2016 Apr;127(4):745-751. doi: 10.1097/AOG.0000000000001359. PMID 27008217
- [Background] Bote ME, Garcia JJ, Hinchado MD, Ortega E. Fibromyalgia: anti-inflammatory and stress responses after acute moderate exercise. PLoS One. 2013 Sep 4;8(9):e74524. doi: 10.1371/journal.pone.0074524. eCollection 2013. PMID 24023948
- [Background] Bottiroli S, Galli F, Viana M, De Icco R, Bitetto V, Allena M, Pazzi S, Sances G, Tassorelli C. Negative Short-Term Outcome of Detoxification Therapy in Chronic Migraine With Medication Overuse Headache: Role for Early Life Traumatic Experiences and Recent Stressful Events. Front Neurol. 2019 Mar 7;10:173. doi: 10.3389/fneur.2019.00173. eCollection 2019. PMID 30899242
- [Background] Bottiroli S, Galli F, Viana M, Sances G, Tassorelli C. Traumatic Experiences, Stressful Events, and Alexithymia in Chronic Migraine With Medication Overuse. Front Psychol. 2018 May 14;9:704. doi: 10.3389/fpsyg.2018.00704. eCollection 2018. PMID 29867669
- [Background] Bottiroli, S., Ghiggia, A., Galli, F., Castelli, L., Guaschino, E., & Tassorelli, C. (2021). Alexithymia and psychological distress in chronic migraine and fibromyalgia: A comparative study. The Journal of Headache and Pain, 132-132.
- [Background] Bottiroli S, Viana M, Sances G, Ghiotto N, Guaschino E, Galli F, Vegni E, Pazzi S, Nappi G, Tassorelli C. Psychological factors associated with failure of detoxification treatment in chronic headache associated with medication overuse. Cephalalgia. 2016 Dec;36(14):1356-1365. doi: 10.1177/0333102416631960. Epub 2016 Feb 15. PMID 26879321
- [Background] Branco JC, Bannwarth B, Failde I, Abello Carbonell J, Blotman F, Spaeth M, Saraiva F, Nacci F, Thomas E, Caubere JP, Le Lay K, Taieb C, Matucci-Cerinic M. Prevalence of fibromyalgia: a survey in five European countries. Semin Arthritis Rheum. 2010 Jun;39(6):448-53. doi: 10.1016/j.semarthrit.2008.12.003. Epub 2009 Feb 27. PMID 19250656
- [Background] Chiarotto A, Viti C, Sulli A, Cutolo M, Testa M, Piscitelli D. Cross-cultural adaptation and validity of the Italian version of the Central Sensitization Inventory. Musculoskelet Sci Pract. 2018 Oct;37:20-28. doi: 10.1016/j.msksp.2018.06.005. Epub 2018 Jun 15. PMID 29966856
- [Background] Cohen ML. Proposed clinical criteria for nociplastic pain in the musculoskeletal system are flawed. Pain. 2022 Apr 1;163(4):e606-e607. doi: 10.1097/j.pain.0000000000002505. No abstract available. PMID 35302978
- [Background] Crofford LJ. Violence, stress, and somatic syndromes. Trauma Violence Abuse. 2007 Jul;8(3):299-313. doi: 10.1177/1524838007303196. PMID 17596347
- [Background] Dahlhamer J, Lucas J, Zelaya C, Nahin R, Mackey S, DeBar L, Kerns R, Von Korff M, Porter L, Helmick C. Prevalence of Chronic Pain and High-Impact Chronic Pain Among Adults - United States, 2016. MMWR Morb Mortal Wkly Rep. 2018 Sep 14;67(36):1001-1006. doi: 10.15585/mmwr.mm6736a2. PMID 30212442
- [Background] de Tommaso M, Sciruicchio V. Migraine and Central Sensitization: Clinical Features, Main Comorbidities and Therapeutic Perspectives. Curr Rheumatol Rev. 2016;12(2):113-26. doi: 10.2174/1573397112666151231110813. PMID 26717950
- [Background] Di Giuseppe M, Perry JC, Lucchesi M, Michelini M, Vitiello S, Piantanida A, Fabiani M, Maffei S, Conversano C. Preliminary Reliability and Validity of the DMRS-SR-30, a Novel Self-Report Measure Based on the Defense Mechanisms Rating Scales. Front Psychiatry. 2020 Aug 26;11:870. doi: 10.3389/fpsyt.2020.00870. eCollection 2020. PMID 33005160
- [Background] Di Tella M, Ghiggia A, Tesio V, Romeo A, Colonna F, Fusaro E, Torta R, Castelli L. Pain experience in Fibromyalgia Syndrome: The role of alexithymia and psychological distress. J Affect Disord. 2017 Jan 15;208:87-93. doi: 10.1016/j.jad.2016.08.080. Epub 2016 Oct 11. PMID 27750065
- [Background] Fayaz A, Croft P, Langford RM, Donaldson LJ, Jones GT. Prevalence of chronic pain in the UK: a systematic review and meta-analysis of population studies. BMJ Open. 2016 Jun 20;6(6):e010364. doi: 10.1136/bmjopen-2015-010364. PMID 27324708
- [Background] Ferrari MD, Klever RR, Terwindt GM, Ayata C, van den Maagdenberg AM. Migraine pathophysiology: lessons from mouse models and human genetics. Lancet Neurol. 2015 Jan;14(1):65-80. doi: 10.1016/S1474-4422(14)70220-0. PMID 25496898
- [Background] Fish RA, McGuire B, Hogan M, Morrison TG, Stewart I. Validation of the chronic pain acceptance questionnaire (CPAQ) in an Internet sample and development and preliminary validation of the CPAQ-8. Pain. 2010 Jun;149(3):435-443. doi: 10.1016/j.pain.2009.12.016. Epub 2010 Feb 25. PMID 20188472
- [Background] Fitzcharles MA, Cohen SP, Clauw DJ, Littlejohn G, Usui C, Hauser W. Nociplastic pain: towards an understanding of prevalent pain conditions. Lancet. 2021 May 29;397(10289):2098-2110. doi: 10.1016/S0140-6736(21)00392-5. PMID 34062144
- [Background] Foster DC, Dworkin RH, Wood RW. Effects of intradermal foot and forearm capsaicin injections in normal and vulvodynia-afflicted women. Pain. 2005 Sep;117(1-2):128-36. doi: 10.1016/j.pain.2005.05.025. PMID 16087295
- [Background] Franke GH, Jaeger S, Glaesmer H, Barkmann C, Petrowski K, Braehler E. Psychometric analysis of the brief symptom inventory 18 (BSI-18) in a representative German sample. BMC Med Res Methodol. 2017 Jan 26;17(1):14. doi: 10.1186/s12874-016-0283-3. PMID 28125960
- [Background] Galli F. Understanding Nociplastic Pain: Building a Bridge between Clinical Psychology and Medicine. J Pers Med. 2023 Feb 10;13(2):310. doi: 10.3390/jpm13020310. PMID 36836544
- [Background] Galli F, Caputi M, Sances G, Vegni E, Bottiroli S, Nappi G, Tassorelli C. Alexithymia in chronic and episodic migraine: a comparative study. J Ment Health. 2017 Jun;26(3):192-196. doi: 10.3109/09638237.2015.1124404. Epub 2016 Jan 6. PMID 26732465
- [Background] Galli F, Tanzilli A, Simonelli A, Tassorelli C, Sances G, Parolin M, Cristofalo P, Gualco I, Lingiardi V. Personality and Personality Disorders in Medication-Overuse Headache: A Controlled Study by SWAP-200. Pain Res Manag. 2019 Jun 12;2019:1874078. doi: 10.1155/2019/1874078. eCollection 2019. PMID 31281555
- [Background] Galvez-Sanchez CM, Duschek S, Reyes Del Paso GA. Psychological impact of fibromyalgia: current perspectives. Psychol Res Behav Manag. 2019 Feb 13;12:117-127. doi: 10.2147/PRBM.S178240. eCollection 2019. PMID 30858740
- [Background] Giesecke J, Reed BD, Haefner HK, Giesecke T, Clauw DJ, Gracely RH. Quantitative sensory testing in vulvodynia patients and increased peripheral pressure pain sensitivity. Obstet Gynecol. 2004 Jul;104(1):126-33. doi: 10.1097/01.AOG.0000129238.49397.4e. PMID 15229011
- [Background] Goadsby PJ, Holland PR, Martins-Oliveira M, Hoffmann J, Schankin C, Akerman S. Pathophysiology of Migraine: A Disorder of Sensory Processing. Physiol Rev. 2017 Apr;97(2):553-622. doi: 10.1152/physrev.00034.2015. PMID 28179394
- [Background] Guidetti V, Galli F, Fabrizi P, Giannantoni AS, Napoli L, Bruni O, Trillo S. Headache and psychiatric comorbidity: clinical aspects and outcome in an 8-year follow-up study. Cephalalgia. 1998 Sep;18(7):455-62. doi: 10.1046/j.1468-2982.1998.1807455.x. PMID 9793697
- [Background] Guma-Uriel L, Penarrubia-Maria MT, Cerda-Lafont M, Cunillera-Puertolas O, Almeda-Ortega J, Fernandez-Vergel R, Garcia-Campayo J, Luciano JV. Impact of IPDE-SQ personality disorders on the healthcare and societal costs of fibromyalgia patients: a cross-sectional study. BMC Fam Pract. 2016 Jun 1;17:61. doi: 10.1186/s12875-016-0464-5. PMID 27245582
- [Background] Harlow BL, Kunitz CG, Nguyen RH, Rydell SA, Turner RM, MacLehose RF. Prevalence of symptoms consistent with a diagnosis of vulvodynia: population-based estimates from 2 geographic regions. Am J Obstet Gynecol. 2014 Jan;210(1):40.e1-8. doi: 10.1016/j.ajog.2013.09.033. Epub 2013 Sep 28. PMID 24080300
- [Background] IASP. International Association for the Study of Pain (IASP) (2017). Terminology; IASP: Washington, DC, USA, 2017.
- [Background] Karsan N, Goadsby PJ. Migraine Is More Than Just Headache: Is the Link to Chronic Fatigue and Mood Disorders Simply Due to Shared Biological Systems? Front Hum Neurosci. 2021 Jun 3;15:646692. doi: 10.3389/fnhum.2021.646692. eCollection 2021. PMID 34149377
- [Background] Katz J, Rosenbloom BN, Fashler S. Chronic Pain, Psychopathology, and DSM-5 Somatic Symptom Disorder. Can J Psychiatry. 2015 Apr;60(4):160-7. doi: 10.1177/070674371506000402. PMID 26174215
- [Background] Kleykamp BA, Ferguson MC, McNicol E, Bixho I, Arnold LM, Edwards RR, Fillingim R, Grol-Prokopczyk H, Turk DC, Dworkin RH. The Prevalence of Psychiatric and Chronic Pain Comorbidities in Fibromyalgia: an ACTTION systematic review. Semin Arthritis Rheum. 2021 Feb;51(1):166-174. doi: 10.1016/j.semarthrit.2020.10.006. Epub 2020 Dec 29. PMID 33383293
- [Background] Lionetti F, Aron A, Aron EN, Burns GL, Jagiellowicz J, Pluess M. Dandelions, tulips and orchids: evidence for the existence of low-sensitive, medium-sensitive and high-sensitive individuals. Transl Psychiatry. 2018 Jan 22;8(1):24. doi: 10.1038/s41398-017-0090-6. PMID 29353876
- [Background] Lumley MA, Krohner S, Marshall LM, Kitts TC, Schubiner H, Yarns BC. Emotional awareness and other emotional processes: implications for the assessment and treatment of chronic pain. Pain Manag. 2021 May;11(3):325-332. doi: 10.2217/pmt-2020-0081. Epub 2021 Feb 3. PMID 33533272
- [Background] Marchi L, Marzetti F, Orru G, Lemmetti S, Miccoli M, Ciacchini R, Hitchcott PK, Bazzicchi L, Gemignani A, Conversano C. Alexithymia and Psychological Distress in Patients With Fibromyalgia and Rheumatic Disease. Front Psychol. 2019 Jul 31;10:1735. doi: 10.3389/fpsyg.2019.01735. eCollection 2019. PMID 31417462
- [Background] Melzack R. The McGill pain questionnaire: from description to measurement. Anesthesiology. 2005 Jul;103(1):199-202. doi: 10.1097/00000542-200507000-00028. PMID 15983473
- [Background] Meston C, Trapnell P. Development and validation of a five-factor sexual satisfaction and distress scale for women: the Sexual Satisfaction Scale for Women (SSS-W). J Sex Med. 2005 Jan;2(1):66-81. doi: 10.1111/j.1743-6109.2005.20107.x. PMID 16422909
- [Background] Modgill G, Jette N, Wang JL, Becker WJ, Patten SB. A population-based longitudinal community study of major depression and migraine. Headache. 2012 Mar;52(3):422-32. doi: 10.1111/j.1526-4610.2011.02036.x. Epub 2011 Nov 15. PMID 22084834
- [Background] Nakamura I, Nishioka K, Usui C, Osada K, Ichibayashi H, Ishida M, Turk DC, Matsumoto Y, Nishioka K. An epidemiologic internet survey of fibromyalgia and chronic pain in Japan. Arthritis Care Res (Hoboken). 2014 Jul;66(7):1093-101. doi: 10.1002/acr.22277. PMID 24403219
- [Background] Naylor, S., Tebbutt, A., & MacPhie, E. (2017). 301. DOING MORE WITH LESS: EVALUATION OF THE CONDENSED FORMAT FIBROMYALGIA EDUCATION GROUP AT THE MINERVA HEALTH CENTRE. Rheumatology, 56(suppl_2).
- [Background] Nijenhuis, E. R., Van der Hart, O., & Kruger, K. (2002). The psychometric characteristics of the Traumatic Experiences Checklist (TEC): First findings among psychiatric outpatients. Clinical Psychology & Psychotherapy: An International Journal of Theory & Practice, 9(3), 200-210.
- [Background] Pergolizzi J, Ahlbeck K, Aldington D, Alon E, Coluzzi F, Dahan A, Huygen F, Kocot-Kepska M, Mangas AC, Mavrocordatos P, Morlion B, Muller-Schwefe G, Nicolaou A, Perez Hernandez C, Sichere P, Schafer M, Varrassi G. The development of chronic pain: physiological CHANGE necessitates a multidisciplinary approach to treatment. Curr Med Res Opin. 2013 Sep;29(9):1127-35. doi: 10.1185/03007995.2013.810615. Epub 2013 Jul 3. PMID 23786498
- [Background] Pukall CF, Goldstein AT, Bergeron S, Foster D, Stein A, Kellogg-Spadt S, Bachmann G. Vulvodynia: Definition, Prevalence, Impact, and Pathophysiological Factors. J Sex Med. 2016 Mar;13(3):291-304. doi: 10.1016/j.jsxm.2015.12.021. PMID 26944461
- [Background] Reed BD, Harlow SD, Sen A, Edwards RM, Chen D, Haefner HK. Relationship between vulvodynia and chronic comorbid pain conditions. Obstet Gynecol. 2012 Jul;120(1):145-51. doi: 10.1097/AOG.0b013e31825957cf. PMID 22914403
- [Background] Rosen R, Brown C, Heiman J, Leiblum S, Meston C, Shabsigh R, Ferguson D, D'Agostino R Jr. The Female Sexual Function Index (FSFI): a multidimensional self-report instrument for the assessment of female sexual function. J Sex Marital Ther. 2000 Apr-Jun;26(2):191-208. doi: 10.1080/009262300278597. PMID 10782451
- [Background] Schweinhardt P, Sauro KM, Bushnell MC. Fibromyalgia: a disorder of the brain? Neuroscientist. 2008 Oct;14(5):415-21. doi: 10.1177/1073858407312521. Epub 2008 Feb 12. PMID 18270311
- [Background] Sluka KA, Clauw DJ. Neurobiology of fibromyalgia and chronic widespread pain. Neuroscience. 2016 Dec 3;338:114-129. doi: 10.1016/j.neuroscience.2016.06.006. Epub 2016 Jun 9. PMID 27291641
- [Background] Sommer C, Hauser W, Burgmer M, Engelhardt R, Gerhold K, Petzke F, Schmidt-Wilcke T, Spath M, Tolle T, Uceyler N, Wang H, Winkelmann A, Thieme K; Arbeitsgemeinschaft der Wissenschaftlichen Medizinischen Fachgesellschaften. [Etiology and pathophysiology of fibromyalgia syndrome]. Schmerz. 2012 Jun;26(3):259-67. doi: 10.1007/s00482-012-1174-0. German. PMID 22760458
- [Background] Stensland SO, Dyb G, Thoresen S, Wentzel-Larsen T, Zwart JA. Potentially traumatic interpersonal events, psychological distress and recurrent headache in a population-based cohort of adolescents: the HUNT study. BMJ Open. 2013 Jul 30;3(7):e002997. doi: 10.1136/bmjopen-2013-002997. PMID 23901028
- [Background] Sutton K, Pukall C, Wild C, Johnsrude I, Chamberlain S. Cognitive, psychophysical, and neural correlates of vulvar pain in primary and secondary provoked vestibulodynia: a pilot study. J Sex Med. 2015 May;12(5):1283-97. doi: 10.1111/jsm.12863. Epub 2015 Mar 23. PMID 25808781
- [Background] Svicher A, Romanazzo S, De Cesaris F, Benemei S, Geppetti P, Cosci F. Mental Pain Questionnaire: An item response theory analysis. J Affect Disord. 2019 Apr 15;249:226-233. doi: 10.1016/j.jad.2019.02.030. Epub 2019 Feb 11. PMID 30776664
- [Background] Tang NK, Beckwith P, Ashworth P. Mental Defeat Is Associated With Suicide Intent in Patients With Chronic Pain. Clin J Pain. 2016 May;32(5):411-9. doi: 10.1097/AJP.0000000000000276. PMID 26201013
- [Background] Thieme K, Mathys M, Turk DC. Evidenced-Based Guidelines on the Treatment of Fibromyalgia Patients: Are They Consistent and If Not, Why Not? Have Effective Psychological Treatments Been Overlooked? J Pain. 2017 Jul;18(7):747-756. doi: 10.1016/j.jpain.2016.12.006. Epub 2016 Dec 27. PMID 28034828
- [Background] Thimm JC, Jordan S, Bach B. The Personality Inventory for DSM-5 Short Form (PID-5-SF): psychometric properties and association with big five traits and pathological beliefs in a Norwegian population. BMC Psychol. 2016 Dec 7;4(1):61. doi: 10.1186/s40359-016-0169-5. PMID 27927237
- [Background] Tietjen GE, Buse DC, Collins SA. Childhood Maltreatment in the Migraine Patient. Curr Treat Options Neurol. 2016 Jul;18(7):31. doi: 10.1007/s11940-016-0415-4. PMID 27194425
- [Background] Tietjen GE, Herial NA, Hardgrove J, Utley C, White L. Migraine comorbidity constellations. Headache. 2007 Jun;47(6):857-65. doi: 10.1111/j.1526-4610.2007.00814.x. PMID 17578536
- [Background] Tsang A, Von Korff M, Lee S, Alonso J, Karam E, Angermeyer MC, Borges GL, Bromet EJ, Demytteneare K, de Girolamo G, de Graaf R, Gureje O, Lepine JP, Haro JM, Levinson D, Oakley Browne MA, Posada-Villa J, Seedat S, Watanabe M. Common chronic pain conditions in developed and developing countries: gender and age differences and comorbidity with depression-anxiety disorders. J Pain. 2008 Oct;9(10):883-91. doi: 10.1016/j.jpain.2008.05.005. Epub 2008 Jul 7. PMID 18602869
- [Background] Uguz F, Cicek E, Salli A, Karahan AY, Albayrak I, Kaya N, Ugurlu H. Axis I and Axis II psychiatric disorders in patients with fibromyalgia. Gen Hosp Psychiatry. 2010 Jan-Feb;32(1):105-7. doi: 10.1016/j.genhosppsych.2009.07.002. Epub 2009 Sep 11. PMID 20114137
- [Background] Van Der Lugt CM, Rollman A, Naeije M, Lobbezoo F, Visscher CM. Social support in chronic pain: development and preliminary psychometric assessment of a new instrument. J Oral Rehabil. 2012 Apr;39(4):270-6. doi: 10.1111/j.1365-2842.2011.02269.x. Epub 2011 Nov 24. PMID 22115492
- [Background] van Middendorp H, Kool MB, van Beugen S, Denollet J, Lumley MA, Geenen R. Prevalence and relevance of Type D personality in fibromyalgia. Gen Hosp Psychiatry. 2016 Mar-Apr;39:66-72. doi: 10.1016/j.genhosppsych.2015.11.006. Epub 2015 Dec 2. PMID 26804772
- [Background] Vos T, Flaxman AD, Naghavi M, Lozano R, Michaud C, Ezzati M, Shibuya K, Salomon JA, Abdalla S, Aboyans V, Abraham J, Ackerman I, Aggarwal R, Ahn SY, Ali MK, Alvarado M, Anderson HR, Anderson LM, Andrews KG, Atkinson C, Baddour LM, Bahalim AN, Barker-Collo S, Barrero LH, Bartels DH, Basanez MG, Baxter A, Bell ML, Benjamin EJ, Bennett D, Bernabe E, Bhalla K, Bhandari B, Bikbov B, Bin Abdulhak A, Birbeck G, Black JA, Blencowe H, Blore JD, Blyth F, Bolliger I, Bonaventure A, Boufous S, Bourne R, Boussinesq M, Braithwaite T, Brayne C, Bridgett L, Brooker S, Brooks P, Brugha TS, Bryan-Hancock C, Bucello C, Buchbinder R, Buckle G, Budke CM, Burch M, Burney P, Burstein R, Calabria B, Campbell B, Canter CE, Carabin H, Carapetis J, Carmona L, Cella C, Charlson F, Chen H, Cheng AT, Chou D, Chugh SS, Coffeng LE, Colan SD, Colquhoun S, Colson KE, Condon J, Connor MD, Cooper LT, Corriere M, Cortinovis M, de Vaccaro KC, Couser W, Cowie BC, Criqui MH, Cross M, Dabhadkar KC, Dahiya M, Dahodwala N, Damsere-Derry J, Danaei G, Davis A, De Leo D, Degenhardt L, Dellavalle R, Delossantos A, Denenberg J, Derrett S, Des Jarlais DC, Dharmaratne SD, Dherani M, Diaz-Torne C, Dolk H, Dorsey ER, Driscoll T, Duber H, Ebel B, Edmond K, Elbaz A, Ali SE, Erskine H, Erwin PJ, Espindola P, Ewoigbokhan SE, Farzadfar F, Feigin V, Felson DT, Ferrari A, Ferri CP, Fevre EM, Finucane MM, Flaxman S, Flood L, Foreman K, Forouzanfar MH, Fowkes FG, Franklin R, Fransen M, Freeman MK, Gabbe BJ, Gabriel SE, Gakidou E, Ganatra HA, Garcia B, Gaspari F, Gillum RF, Gmel G, Gosselin R, Grainger R, Groeger J, Guillemin F, Gunnell D, Gupta R, Haagsma J, Hagan H, Halasa YA, Hall W, Haring D, Haro JM, Harrison JE, Havmoeller R, Hay RJ, Higashi H, Hill C, Hoen B, Hoffman H, Hotez PJ, Hoy D, Huang JJ, Ibeanusi SE, Jacobsen KH, James SL, Jarvis D, Jasrasaria R, Jayaraman S, Johns N, Jonas JB, Karthikeyan G, Kassebaum N, Kawakami N, Keren A, Khoo JP, King CH, Knowlton LM, Kobusingye O, Koranteng A, Krishnamurthi R, Lalloo R, Laslett LL, Lathlean T, Leasher JL, Lee YY, Leigh J, Lim SS, Limb E, Lin JK, Lipnick M, Lipshultz SE, Liu W, Loane M, Ohno SL, Lyons R, Ma J, Mabweijano J, MacIntyre MF, Malekzadeh R, Mallinger L, Manivannan S, Marcenes W, March L, Margolis DJ, Marks GB, Marks R, Matsumori A, Matzopoulos R, Mayosi BM, McAnulty JH, McDermott MM, McGill N, McGrath J, Medina-Mora ME, Meltzer M, Mensah GA, Merriman TR, Meyer AC, Miglioli V, Miller M, Miller TR, Mitchell PB, Mocumbi AO, Moffitt TE, Mokdad AA, Monasta L, Montico M, Moradi-Lakeh M, Moran A, Morawska L, Mori R, Murdoch ME, Mwaniki MK, Naidoo K, Nair MN, Naldi L, Narayan KM, Nelson PK, Nelson RG, Nevitt MC, Newton CR, Nolte S, Norman P, Norman R, O'Donnell M, O'Hanlon S, Olives C, Omer SB, Ortblad K, Osborne R, Ozgediz D, Page A, Pahari B, Pandian JD, Rivero AP, Patten SB, Pearce N, Padilla RP, Perez-Ruiz F, Perico N, Pesudovs K, Phillips D, Phillips MR, Pierce K, Pion S, Polanczyk GV, Polinder S, Pope CA 3rd, Popova S, Porrini E, Pourmalek F, Prince M, Pullan RL, Ramaiah KD, Ranganathan D, Razavi H, Regan M, Rehm JT, Rein DB, Remuzzi G, Richardson K, Rivara FP, Roberts T, Robinson C, De Leon FR, Ronfani L, Room R, Rosenfeld LC, Rushton L, Sacco RL, Saha S, Sampson U, Sanchez-Riera L, Sanman E, Schwebel DC, Scott JG, Segui-Gomez M, Shahraz S, Shepard DS, Shin H, Shivakoti R, Singh D, Singh GM, Singh JA, Singleton J, Sleet DA, Sliwa K, Smith E, Smith JL, Stapelberg NJ, Steer A, Steiner T, Stolk WA, Stovner LJ, Sudfeld C, Syed S, Tamburlini G, Tavakkoli M, Taylor HR, Taylor JA, Taylor WJ, Thomas B, Thomson WM, Thurston GD, Tleyjeh IM, Tonelli M, Towbin JA, Truelsen T, Tsilimbaris MK, Ubeda C, Undurraga EA, van der Werf MJ, van Os J, Vavilala MS, Venketasubramanian N, Wang M, Wang W, Watt K, Weatherall DJ, Weinstock MA, Weintraub R, Weisskopf MG, Weissman MM, White RA, Whiteford H, Wiersma ST, Wilkinson JD, Williams HC, Williams SR, Witt E, Wolfe F, Woolf AD, Wulf S, Yeh PH, Zaidi AK, Zheng ZJ, Zonies D, Lopez AD, Murray CJ, AlMazroa MA, Memish ZA. Years lived with disability (YLDs) for 1160 sequelae of 289 diseases and injuries 1990-2010: a systematic analysis for the Global Burden of Disease Study 2010. Lancet. 2012 Dec 15;380(9859):2163-96. doi: 10.1016/S0140-6736(12)61729-2. PMID 23245607
- [Background] Wesselmann U, Bonham A, Foster D. Vulvodynia: Current state of the biological science. Pain. 2014 Sep;155(9):1696-1701. doi: 10.1016/j.pain.2014.05.010. Epub 2014 May 22. No abstract available. PMID 24858303
- [Background] Westergaard ML, Hansen EH, Glumer C, Jensen RH. Prescription pain medications and chronic headache in Denmark: implications for preventing medication overuse. Eur J Clin Pharmacol. 2015 Jul;71(7):851-60. doi: 10.1007/s00228-015-1858-3. Epub 2015 May 14. PMID 25967539
- [Background] Wolfe F, Clauw DJ, Fitzcharles MA, Goldenberg DL, Hauser W, Katz RL, Mease PJ, Russell AS, Russell IJ, Walitt B. 2016 Revisions to the 2010/2011 fibromyalgia diagnostic criteria. Semin Arthritis Rheum. 2016 Dec;46(3):319-329. doi: 10.1016/j.semarthrit.2016.08.012. Epub 2016 Aug 30. PMID 27916278
- [Result] Aaron RV, Finan PH, Wegener ST, Keefe FJ, Lumley MA. Emotion regulation as a transdiagnostic factor underlying co-occurring chronic pain and problematic opioid use. Am Psychol. 2020 Sep;75(6):796-810. doi: 10.1037/amp0000678. PMID 32915024

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-10-26): https://cdn.clinicaltrials.gov/large-docs/71/NCT06138171/Prot_SAP_000.pdf
  • Informed Consent Form (2023-09-12): https://cdn.clinicaltrials.gov/large-docs/71/NCT06138171/ICF_001.pdf